CLINICAL TRIAL: NCT00566436
Title: The Surgical Treatment of Long Occlusions of the Superficial Femoral Artery: Initial Success and Long Term Results of Remote Endarterectomy Versus Suprageniculate Bypass Surgery
Brief Title: Remote Endarterectomy Versus Suprageniculate Femoropopliteal Bypass
Acronym: REVAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Antonius Hospital (Other)
Collaborators: UMC Utrecht (Other); Albert Schweitzer Hospital, Netherlands (Unknown); Amphia Hospital (Other)
Responsible Party: Drs SS Gisbertz, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-04.04; P.04.1298L
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2007-11

CONDITIONS: Peripheral Arterial Occlusive Disease; Atherosclerosis
Keywords: Peripheral Arterial Occlusive Disease; Superficial Femoral Artery; Remote Endarterectomy; Suprageniculate Bypass Surgery; Blood Vessel Prosthesis Implantation; Vascular Patency
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- REA (Active Comparator): Patients presenting with a long occlusion of the superficial femoral artery enrolled in REA arm will undergo remote endarterectomy of the occluded superficial femoral artery
  Interventions: Procedure: Remote endarterectomy of the superficial femoral artery
- Bypass (Active Comparator): Patients presenting with a long occlusion of the superficial femoral artery enrolled in Bypass arm will undergo suprageniculate femoropopliteal bypass surgery to bypass the occluded superficial femoral artery
  Interventions: Procedure: Suprageniculate femoropopliteal bypass

INTERVENTIONS:
Procedure: Remote endarterectomy of the superficial femoral artery — Exposure of the common femoral, superficial femoral and profunda femoral artery through a single groin incision. Arteriotomy in the proximal SFA followed by dissection of the intima core beyond the occluded segment using the Vollmar ringstripper. The ringstripper is exchanged for a Mollring cutter all under fluoroscopic guidance. With the Mollring Cutter transection of intima core is carried out, remote from the site of entry. After removal of the intima core the transection zone is secured with an aSpire stent after balloon angioplasty. A completion arteriography will verify a patent artery, and embolectomy can be performed when necessary. As indicated a common femoral artery and profundaplasty can be performed and the arteriotomy may be closed with or without patch.
  Other Names: Remote superficial artery endarterectomy; Distal cutting endarterectomy
  Arms: REA
Procedure: Suprageniculate femoropopliteal bypass — Groin and suprageniculate incision, venous (Saphenous vein) or PTFE graft with end to side anastomoses. If the saphenous vein is truly applicable for grafting will ultimately be an intra-operative decision (despite pre-operative venous mapping)
  Other Names: Above knee bypass; Femoropopliteal bypass
  Arms: Bypass

SUMMARY:
The objective of this study is to compare remote superficial femoral artery endarterectomy with suprageniculate bypass surgery in the treatment of long occlusions of the superficial femoral artery. The study hypothesis is that patency rates are comparable and therefore the minimal invasive remote superficial femoral artery endarterectomy can be considered in patients presenting with a long occlusion of the superficial femoral artery.

DETAILED DESCRIPTION:
Different strategies exist in the treatment of chronic long occlusions of the superficial femoral artery and yet we still suffer a significant percentage of restenosis, re-occlusions and even major amputations, reason for continuous development of new techniques. One such technique is the recently developed minimal invasive remote endarterectomy, which shows promising patency rates and possibly less complications with earlier recovery. A more experienced and the most implemented technique is the suprageniculate femoropopliteal bypass graft, which, when using the saphenous vein, has proved durable. A randomized trial comparing both modalities was lacking so far, what makes the objective of this study a comparison of patency rates between those 2 techniques in a randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with Fontaine IIB, III, IV ischemia
* Long (>10 cm) occlusion of the superficial femoral artery, with patent popliteal artery and at least 1 patent crural vessel
* Atherosclerotic disease

Exclusion Criteria:

* Previous operations on the superficial femoral artery
* Radiation therapy groin/leg region
* Diameter superficial femoral artery < 4 mm
* Contrast allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2004-10; Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
(re-)occlusion of the endarterectomized superficial femoral artery or suprageniculate femoropopliteal bypass | 5 year

SECONDARY OUTCOMES:
(a)symptomatic (re)stenosis of the superficial femoral artery or bypass for which a re-intervention was carried out | 5 year
major amputation of the ipsilateral leg | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne S Gisbertz, MD, Principal Investigator — St. Antonius Hospital; Jean Paul PM de Vries, MD, PhD, Principal Investigator — St. Antonius Hospital; Frans L Moll, MD, PhD, Principal Investigator — UMC Utrecht
Locations (4):
- Netherlands (4):
  - Amphia Hospital, Breda, North Brabant
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - St Antonius Hospital, Nieuwegein, Utrecht
  - UMC Utrecht, Utrecht, Utrecht

REFERENCES:
- [Background] Smeets L, Ho GH, Hagenaars T, van den Berg JC, Teijink JA, Moll FL. Remote endarterectomy: first choice in surgical treatment of long segmental SFA occlusive disease? Eur J Vasc Endovasc Surg. 2003 Jun;25(6):583-9. doi: 10.1053/ejvs.2002.1921. PMID 12787704
- [Derived] Gisbertz SS, Ramzan M, Tutein Nolthenius RP, van der Laan L, Overtoom TT, Moll FL, de Vries JP. Short-term results of a randomized trial comparing remote endarterectomy and supragenicular bypass surgery for long occlusions of the superficial femoral artery [the REVAS trial]. Eur J Vasc Endovasc Surg. 2009 Jan;37(1):68-76. doi: 10.1016/j.ejvs.2008.09.014. Epub 2008 Nov 5. PMID 18990592